CLINICAL TRIAL: NCT06471504
Title: Use of Eye Tracking to Aid in Autism Risk Detection
Acronym: RCFET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Rebecca McNally Keehn, Assistant Professor of Pediatrics, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21697
Record Dates: First submitted 2024-05-24; First posted 2024-06-24 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-03

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Children Undergoing Developmental Evaluation (Experimental): Children undergoing a standard of care developmental evaluation will be enrolled into the study. After the completion of the developmental evaluation, research participation includes a one-time eye-tracking activity in which the child will view a series of different pictures and movies while their eye movements are tracked and recorded.
  Interventions: Diagnostic Test: Eyelink Portable Duo

INTERVENTIONS:
Diagnostic Test: Eyelink Portable Duo — Eye-tracking data will be collected using a commercially-available remote eye-tracking system (Eyelink Portable Duo). Eye movements and pupil diameter will be collected while participants view a series of developmentally appropriate pictures and movies. The eye-tracker consists of two cameras; one that monitors eye movements and a second scene camera that monitors head movements, which permits eye tracking to take place without any equipment touching the child. Children will be asked to sit in highchair or on their caregiver's lap and will face a computer monitor. After a sticker is applied to the child's forehead and brief eye-movement calibration completed, next visual stimuli (i.e., pictures and videos) will be presented on a laptop computer monitor that is placed at approximately 60-80cm from the child. The eye tracking portion of the visit will last approximately 15 minutes or until the child is no longer able to attend to pictures/videos.

SUMMARY:
The study will use a non-invasive remote eye-tracking system (Eyelink Portable Duo) to acquire a short series of eye-tracking measures.

DETAILED DESCRIPTION:
The study will use a non-invasive remote eye-tracking system (Eyelink Portable Duo) to acquire a short series (less than 15 mins) of eye-tracking measures (e.g., looking time, pupil diameter, oculomotor dynamics), which may be associated with autism in young children ages 12-48 months. We will recruit children from Riley Hospital for Children at Indiana University Health clinics to determine whether these measures may help determine autism risk.

ELIGIBILITY:
Inclusion Criteria:

* Young children ages 12-48 months scheduled for health care visits at Riley Hospital for Children at Indiana University Health clinics (e.g., Pediatric Care Center clinics).
* Children must have English- or Spanish-speaking caregivers.
* Children must have a legal guardian that is able to provide consent.

Exclusion Criteria:

* Child is younger than 12 months or older than 48 months.
* Child's caregiver(s) is not English- or Spanish-speaking.

Ages: 12 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Agreement between eye-tracking biomarker score and diagnosis | Day 1
  The composite eye-tracking biomarker score, a consolidated measure based on eye-tracking indices that predict autism outcome, will be compared to the categorical autism diagnosis (autism presence/absence). Clinical diagnosis is obtained based upon a standard clinical evaluation conducted by an expert clinical psychologist. The evaluation will include 1) a semi-structured caregiver(s) clinical interview to gather information about developmental history and autism symptoms and 2) a battery of standardized child clinical observational measures. The evaluation will be conducted over a one-time 2-hour clinical autism evaluation. Eye-tracking will be recorded immediately following the clinical evaluation for a period of up to 15 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca R McNally Keehn, PhD, HSPP, Principal Investigator — IU School of Medicine
Locations (1):
- Riley Hospital for Children, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No